CLINICAL TRIAL: NCT05585073
Title: Factors Affecting the Difficulty of Laparoscopic D2 Lymph Node Dissection for Gastric Cancer:a Retrospective Cohort Study
Brief Title: Factors Affecting the Difficulty of Laparoscopic D2 Lymph Node Dissection for Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Clinical Professor, Fujian Medical University
Other Study IDs: SD-GC
Record Dates: First submitted 2022-10-15; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Surgery-Complications
MeSH Terms: interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- qualified of D2 Lymph node dissection group
  Interventions: Other: Whether lymph node dissection is qualified or not
- not-qualified D2 Lymph node dissection group
  Interventions: Other: Whether lymph node dissection is qualified or not

INTERVENTIONS:
Other: Whether lymph node dissection is qualified or not — Klass-02-QC LND scale and general error score tool were used to quantitatively evaluate the intraoperative performance of D2 LND

SUMMARY:
Laparoscopic D2 lymph node dissection (LND) for gastric cancer has a wide range of operations and a high degree of difficulty.The purpose of this study was to evaluate the relationship between clinicopathological factors and the difficulty of laparoscopic D2 LND.

ELIGIBILITY:
Inclusion Criteria:

1. all patients undergoing laparoscopic surgery
2. Laparoscopic system is 2D and has complete D2 lymph node dissection.

Exclusion Criteria:

1. patients undergoing laparotomy
2. incomplete video or clinicopathological information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The CLASS-01 trial is a prospective multicenter randomized controlled study (ClinicalTrials.gov.number:NCT01609309) to compare the oncological efficacy of laparoscopy and laparotomy in the treatment of locally advanced distal gastric cancer. In this study, 119 patients who underwent laparoscopic surgery at our center who participated in CLASS-01 were selected. All the patients were operated with 2D laparoscopic system.The 2D/3D trial is a prospective clinical trial (ClinicalTrials.gov.number:NCT02327481) that compares the curative effect of 2D and 3D laparoscopic radical gastrectomy in our center. Seventy cases of 2D laparoscopic distal gastrectomy (LDG) were selected
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
surgery complicated | 30 days after operation
  Incidence of operative complications between qualified group and unqualified group

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastric Surgery, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lu J, Huang JB, Wu D, Xie JW, Wang JB, Lin JX, Zheng CH, Huang CM, Li P. Factors affecting the quality of laparoscopic D2 lymph node dissection for gastric cancer: a cohort study from two randomized controlled trials. Int J Surg. 2023 May 1;109(5):1249-1256. doi: 10.1097/JS9.0000000000000290. PMID 37026819